CLINICAL TRIAL: NCT00928928
Title: Study of the Oxidative Stress in Patients With Colorectal Cancer. Open vs Laparoscopic Approach
Brief Title: Oxidative Stress Markers in Open and Laparoscopic Colectomy for Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: G. Hatzikosta General Hospital (Other)
Collaborators: University of Ioannina (Other)
Responsible Party: George Pappas-Gogos,MD, G Hatzikosta General Hospital, Ioannina, Greece
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: GH-1948-03; GHDS-12345-3
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Last update posted 2009-06-26 (Estimated); Status verified 2009-06

CONDITIONS: Colorectal Cancer
Keywords: Lipid peroxidation; Protein peroxidation; DNA peroxidation; RNA peroxidation; Cytokines; hsCRP; Oxidative stress markers; Open surgery; Laparoscopic surgery
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Open group (Active Comparator): Group of patients operated with open approach for colorectal cancer
  Interventions: Procedure: Open colectomy
- laparoscopic group (Active Comparator): Group of patients operated with laparoscopic approach for colorectal cancer
  Interventions: Procedure: laparoscopic colectomy

INTERVENTIONS:
Procedure: Open colectomy — Open colectomy. Epidural anaesthesia used
  Arms: Open group
Procedure: laparoscopic colectomy — Laparoscopic colectomy. Epidural anaesthesia used
  Arms: laparoscopic group

SUMMARY:
Contribution to the study of oxidative stress markers in laparoscopic vs open colectomy for colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

* colorectal cancer

Exclusion Criteria:

* metastases
* recurrent disease
* chronic diseases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-01; Primary Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Oxidative stress markers in patients with colorectal cancer operated with open or laparoscopic approach | preoperative, intraoperative, 6h postop, 24h postop

CONTACTS AND LOCATIONS:
Locations (1):
- G Hatzikosta General Hospital, Ioannina, Greece

REFERENCES:
- [Derived] Pappas-Gogos G, Tellis C, Lasithiotakis K, Tselepis AD, Tsimogiannis K, Tsimoyiannis E, Chalkiadakis G, Chrysos E. Oxidative stress markers in laparoscopic versus open colectomy for cancer: a double-blind randomized study. Surg Endosc. 2013 Jul;27(7):2357-65. doi: 10.1007/s00464-013-2788-8. Epub 2013 Feb 13. PMID 23404145